CLINICAL TRIAL: NCT06731439
Title: Does Starting Feeds on the First Day of Life Help Premature Infants Reach Full Volume Feeds Sooner?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-09828-FB
Record Dates: First submitted 2024-07-22; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Extra Uterine Growth Restriction; Premature Infant Disease; VLBW - Very Low Birth Weight Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early feeding arm (Experimental)
  Interventions: Other: Starting feeds within 6 hours of life
- Control arm (Active Comparator)
  Interventions: Other: Standard feeding protocol

INTERVENTIONS:
Other: Starting feeds within 6 hours of life — Starting feeds within 6 hours of life
  Arms: Early feeding arm
Other: Standard feeding protocol — Starting feeds based on standard protocol as per primary team
  Arms: Control arm

SUMMARY:
Feeding advancements in ELBW infants have evolved over decades. The fear of causing mortality and morbidity, notably NEC, have made providers cautious when advancing feeds. ELBW infants initially remained NPO for several days before initiating trophic feeds. However, data then showed that there was no increase in mortality and morbidity if trophic feeds were initiated earlier. Then data showed that a short duration of trophic feeds did not increase mortality and morbidity when compared to a prolonged duration. More recent data showed that enteral feeding should be initiated early, preferably within 24 hours of birth, because it may promote feeding tolerance, shorten the time to reach total enteral feeding, and reduce the incidence of extrauterine growth restriction and late onset sepsis without increasing the risk of developing NEC. The management of enteral nutrition in ELBW infants is still very variable. For example, there is no consensus on the optimal time point after birth at which enteral nutrition can be started. This study evaluates the benefits of starting feeds by 6 hours of life Purpose: The primary aim of this study is to evaluate if in infants ≤ 1000g birth weight, is there a benefit initiating feeds by 6 hours of life (compared to current feeding practice data of 3 days of life) on decreasing the time to attain full feeds in the first 30 days of life. The secondary aim is to evaluate if antenatal feeding discussions would streamline feeding management post-delivery.

DETAILED DESCRIPTION:
Rationale: Although current evidence supports initiating enteral feedings as early as the first day of life in extremely low birth weight infants, there are two main barriers that are usually associated with the initiation of feeding not taking place until an average of the third day of life. Since it is common to supplement the infant's nutrition with donor breast milk, and since donor breast milk requires parental consent, the process of consenting is usually done after the infant is born. This would be the time when the parents are updated with the status of their child and the time when other consents are taken. For example, this would be the time to talk about and take consent for blood transfusions, central line placement, and donor breast milk supplementing the infant's nutrition. The mother is the one most commonly giving consent. In situations after cesarean section or after receiving pain medications, the mother is not in a state where she can be approached for consent. This is typically not an issue for interventions like blood transfusions and central line insertions as the need does not arise typically until after a few days. However, when it comes to enteral feeding, it is recommended to start feeding as early as possible. However, because of the previously listed reasons, this sometimes gets pushed further until the mother is in a more stable situation to approach her for consent.

Another important aspect of feeding pertains to what is considered feeding and what is considered gut priming. It is generally considered that enteral feedings of 10 ml/kg/day are not enough volume to be considered "feeding." This volume is considered more of gut priming that stimulates gut enzymes to get produced and starts the clock for the eventual advancement of feeds. For these initial 10 ml/kg/day volume feeds, the term minimal enteral nutrition has been commonly used. In patients to be enrolled in this study, this will come out to be an average of 0.75 ml every 3 hours, a volume that is typically less than the volume of gastric juice being internally produced by the infant. It is also a volume so small that it is not thought to lead to any significant negative sequelae.

On the other hand, research has shown that prolonged enteral fasting may diminish the functional adaptation of the immature gastrointestinal tract and extend the need for parenteral nutrition along with its risk of sepsis-related morbidity and mortality. Research has also shown that the initiation of early enteral feeds could release trophic endogenous agents and inhibit the release of inflammatory mediators and cytokines. It also assists with the development of the intestinal mucosa, activates digestive enzymes, and improves digestion and absorption to avoid the complications associated with vascular catheterization, sepsis, long-term fasting, and vascular alimentation.

There are no uniform guidelines of how fast to advance feeds in this premature infant population. Depending on the practice, it may take a premature infant 7-15 days to reach the 150 ml/kg/day target volume.

Starting feeds by 6 hours is expected to initiate the feeding process for premature infants and be associated with several benefits. The aim of this study is to investigate if finalizing nutritional care plans with the mother antenatally offers any clinically beneficial outcomes in either streamlining the nutritional care plan as a short-term outcome or being associated with beneficial long-term outcomes. This is currently not practiced because either there is not enough personnel or it is felt not of a high yield because the mother may not end up delivering and come back at another visit to deliver. The study would leverage that starting feeds by 6 hours of life is not considered unsafe because the volume of milk that would be given every 3 hours is <1ml. However, starting early would have helped the infant start the feeding advancement process. The focus is more on "starting" than on "feeding" since the volume received in the first 24 hours is not considered food as much as it is considered gut priming. In other words, the treatment arm group that will have their feeds started by 6 hours of age will have the benefit of having their nutrition clock started earlier when compared to the current standard of care.

Study Project Population:

Infants will be eligible for the study if they have a birth weight ≤1000g and are born in the Regional One Health neonatal intensive care unit in Memphis, TN, during study enrollment. In addition, the clinical care team at the time of enrollment must agree with the neonate's participation. Infants found to have congenital malformations, congenital gastrointestinal obstructions, on more than one pressor, or on dopamine > 5 mcg/kg/min will be excluded. Infants clinically progressing towards imminent death will also be excluded. The mothers of these infants will also be included as part of the study population as the investigators will be collecting maternal health information as it directly affects the neonates.

Research Design:

This will be a prospective randomized controlled trial. The study will be unblinded and conducted at Regional One Health. The target population will be infants with a birth weight of ≤1000g. After informed consent is obtained from parents and after birth but before 6 hours of life, infants meeting the criteria will be randomized to one of two arms: early feeding (intervention group) or standard protocol feeding (control group). In the intervention group, feeds of expressed breast milk, donor breast milk, or formula will be initiated within 6 hours of life based on the mother's feeding preference obtained during the antenatal consent. Feeds will be advanced daily (10 ml/kg/day in the <750g birth weight group and 15 ml/kg/day in the 751-1000g birth weight group) and managed by the primary care team based on their assessment. In the control group, the primary care team will start feedings based on the current protocol. This includes not advancing for the first three days after feeding initiation for infants weighing < 750g per current feeding protocol. If randomized to the control group, all feeding management initiation, advancement, and obtaining consent for donor breast milk will be done by the primary care team. This step is important as it helps to evaluate if antenatal feeding discussions would streamline feeding management post-delivery.

Study Project/Procedure: The growth indices , including height (cm), weight (g), head circumference (cm), and calculated BMI (kg/m2), will be performed weekly as part of our unit's standard practice for all infants admitted. Patient data will be collected from medical records at regular intervals during the study. The primary medical team will manage all medical and feeding-related decisions. The maternal data that the investigators will be collecting for this study from the mother's chart is information such as age, BMI, medications used during pregnancy, medical problems such as diabetes or high blood pressure, and other information that could directly influence the neonate. Milk fortification will take place when feeding volumes reach 40 ml/kg/d. All patients will have feedings temporarily stopped during blood transfusions as per unit guidelines. The primary team can decide on feeding advancement if they plan to administer more than 48 hours of antibiotics. The volume used to start the feeding is not large enough to likely be associated with any feeding intolerance. In both the treatment and control groups, if the primary team decides that the infant is not tolerating feeding, then standard clinical interventions are applicable. These could range from decreasing the volume of feeding to a lower volume or even stopping the feeds completely. Feeding intolerance is not uncommon in this population and both interventions of either decreasing the volume or stopping the feeding are also common interventions. If feeding advancements are paused or feedings are stopped altogether, the primary team will be asked to document their concerns and reasons why feedings are paused or stopped. This will be evaluated every 12 hours.

At a Power=80%, α=5%, and to detect a mean difference of 4(±5) days between the early feeding intervention group and the control group to reach full feeds, a sample size of 52 in each arm is required. The investigators expect to recruit 104 infants in less than 2 years based on current admission rates. With an additional 20% for replacements, a total of 124 infants or 248 infant-mother pairs.

Subjects will participate in the study until hospital discharge.

Outcome Measures: The primary objective of this study is to evaluate if early feeding started at 6 hours of age shortens the time to attain full feeds in the first 30 days of life when compared to starting feeds based on current ROH standard protocol.

Secondary outcomes to be assessed from date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 20 weeks of age will include:

1. Days to goal enteral feeds (days)
2. Days of central line use (days)
3. Days of TPN use (days)
4. Number of feeding intolerance events(feedings held for >24 hours per clinician judgment due to gastrointestinal symptoms such as emesis, abdominal distention, etc.) (N)
5. Time to regain birth weight) (days)
6. anthropometric parameters at birth, at 1500 g weight mark, at 36 weeks postmenstrual age, and at discharge: weight (grams), length (cm), and head circumference (cm)
7. Bronchopulmonary dysplasia development assessed at 36 weeks postmenstrual age (Y/N)
8. IVH grade (I to IV) assessed at 2 weeks and 4 weeks of age (severe defined as Grade III and Grade IV (Y/N))
9. Days on antibiotics (days) during the entire hospitalization from birth until discharge
10. Length of NICU stay (days) from birth until discharge
11. The presence of a patent ductus arteriosus incidence requiring treatment anytime from birth until discharge (Y/N)

10- Necrotizing enterocolitis incidence requiring treatment anytime from birth until discharge (Y/N) 11- Catheter-related infections anytime from birth until discharge (Y/N) 10- Death incidence (Y/N) 12-Number of subjects not consented and the reason from the study's first enrollment date until study closure.

ELIGIBILITY:
Inclusion Criteria:

1. All infants less than or equal to 1000 g
2. Clinical care team in agreement with patient's participation
3. All mothers with pregnancies with EFW close to 1000g or less.

Exclusion Criteria:

1 congenital malformations that may affect gastro intestinal perfusion

2 Clinically progressing towards imminent death

3 congenital gastrointestinal obstructions

4 Mothers unlikely to deliver infants ≤ 1000g

5 Infant on pressors other than dopamine given at < 5mcg/kg/min. Dopamine is an exclusion if administered at a dose exceeding 5mcg/kg/min.

6 Mothers who are not in a sound mental state to be consented either to their critical condition, intubated, sedated, for examples

7 Mothers who are critically ill where by it is felt that mom will not be able to participate in the consent

Ages: 1 Minute to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Day of life reaching full feeds | From birth until day of life full feeds reached in the first 30 days of life
  The primary outcome is the age in days in the first 30 days of life when the infant reaches full feeds.

SECONDARY OUTCOMES:
Secondary Outcomes | From birth until hospital discharge
  Days of central line use (Days)
Secondary Outcomes | From birth until hospital discharge
  Days of TPN use (Days)
Secondary Outcomes | From birth until 30 days of life
  The number of feeding intolerance events defined as feedings held for >24 hours per clinician judgment due to gastrointestinal symptoms such as emesis, abdominal distention, etc.
Secondary Outcomes | From birth until hospital discharge
  The development of BPD (Y/N)
Secondary Outcomes | From birth until hospital discharge
  The development of IVH (Y/N)
Secondary Outcomes | From birth until hospital discharge
  Days of antibiotic use (Days)
Secondary Outcomes | From birth until hospital discharge
  Length of NICU stay (Days)
Secondary Outcomes | From birth until hospital discharge
  PDA incidence requiring treatment (Y/N)
Secondary Outcomes | From birth until hospital discharge
  The development of CLABSI (Y/N)
Secondary Outcomes | From birth until hospital discharge
  The development of Death (Y/N)
Secondary Outcomes | From birth until hospital discharge
  The development of NEC (Y/N)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Elabiad, MD, Principal Investigator — UTHSC
Locations (1):
- Regional One Health, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker LA, Desorcy-Scherer K, Magalhaes M. Feeding Strategies in Preterm Very Low Birth-Weight Infants: State-of-the-Science Review. Adv Neonatal Care. 2021 Dec 1;21(6):493-502. doi: 10.1097/ANC.0000000000000849. PMID 33675303
- [Background] Walsh V, Brown JVE, Copperthwaite BR, Oddie SJ, McGuire W. Early full enteral feeding for preterm or low birth weight infants. Cochrane Database Syst Rev. 2020 Dec 27;12(12):CD013542. doi: 10.1002/14651858.CD013542.pub2. PMID 33368149
- [Background] Morgan J, Bombell S, McGuire W. Early trophic feeding versus enteral fasting for very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD000504. doi: 10.1002/14651858.CD000504.pub4. PMID 23543508
- [Background] Gao L, Shen W, Wu F, Mao J, Liu L, Chang YM, Zhang R, Ye XZ, Qiu YP, Ma L, Cheng R, Wu H, Chen DM, Chen L, Xu P, Mei H, Wang SN, Xu FL, Ju R, Zheng Z, Lin XZ, Tong XM; Chinese Multicenter EUGR Collaborative Group. Effect of early initiation of enteral nutrition on short-term clinical outcomes of very premature infants: A national multicenter cohort study in China. Nutrition. 2023 Mar;107:111912. doi: 10.1016/j.nut.2022.111912. Epub 2022 Nov 12. PMID 36577163